CLINICAL TRIAL: NCT02924493
Title: Dietary Treatment of Endometriosis-related Irritable Bowel Syndrome: A Pilot Study
Brief Title: Dietary Treatment of Endometriosis-related Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Diet-in-endometriosis
Record Dates: First submitted 2016-09-15; First posted 2016-10-05 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2017-10

CONDITIONS: Endometriosis; Irritable Bowel Syndrome; Visceral Syndrome; Visceral Hypersensitivity
Keywords: Endometriosis; IBS; Irritable bowel syndrome; low FODMAP diet; FODMAPs; visceral syndrome; fermentable carbohydrates; visceral hypersensitivity; cross organ effect
MeSH Terms: conditions — Endometriosis; Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low FODMAP diet (Experimental): This group will follow a exclusion diet called low FODMAP diet, which is a diet with restriction of fermentable carbohydrates. The patients will be guided on how to avoid some foods and how to include others. The patients will follow the diet for four weeks.
  Interventions: Other: Diet low in fermentable carbohydrates (low FODMAP diet)
- Control diet (Placebo Comparator): This group will follow a placebo diet, which is designed to imitate the low FODMAP diet by restricting specific foods. However, it is randomly selected foods that will be excluded in this diet, so that it works only as a control diet. The patients in this group will also be guided how to follow the diet for four weeks.
  Interventions: Other: Diet low in fermentable carbohydrates (low FODMAP diet)

INTERVENTIONS:
Other: Diet low in fermentable carbohydrates (low FODMAP diet) — The participants follow the diet in 4 weeks. They have been provided with some foods (bread, pasta, cereal products), but will by the rest themselves. They have been provided with lists of foods to include and foods to avoid. They have also been provided with suggestions to a 4 week meal plan, based in their individual need for energy.

SUMMARY:
Many patients with endometriosis experience extra genital and abdominal symptoms as a major part of their problem. This includes gastrointestinal dysfunction with pain, urinary symptoms compatible with interstitial cystitis and gastrointestinal symptoms resembling the irritable bowel syndrome (IBS). Such problems may be secondary to changes in autonomous neuronal structure and function elicited by the endometriotic elements, which may cause a "visceral syndrome" with the above mentioned symptoms.

The investigators hypothesize that dietary treatment will improve the experience of gastrointestinal symptoms, pain and quality of life in patients with endometriosis-related irritable bowel syndrome. The aim of this first randomized, placebo controlled pilot study investigating patients with both endometriosis and IBS, is to test the application of a low FODMAP diet and a placebo diet for endometriosis-related IBS-like symptoms in order to stablish a platform for a randomized controlled study. Thus, the primary aim of this pilot study is to investigate the applicability of a placebo diet in patients with endometriosis and to investigate the compliance in both intervention group and control group. In addition, the aim is to investigate whether the participants find the diet manageable and whether they are able to identify the placebo diet.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 18-50 years
* Fluid spoken and written Danish
* Diagnosed endometriosis (laparoscopy and/or MR-scan) at least one year ago and sufficient treated regarding medicine and surgery. Participant will be asked to bring a copy of their medical record from the hospital or from www.sundhed.dk to verify the diagnosis.
* Diagnosis of irritable bowel syndrome according to the Rome III criteria. Both previous diagnosis and undiagnosed patients are included, as long as the study group evaluates that the patient meets the Rome III criteria.
* Accept to follow a controlled exclusion diet for all meals for four weeks with only few accepted deviations from the diet.

Exclusion Criteria:

* Premature menopause
* Organic bowel disease (Celiac disease, IBD, bowel endometriosis, malignant disease)
* New therapeutic interventions during study period (medical/lifestyle/psychological). Already ongoing treatment is accepted.
* Psychiatric disorder, psychotropic drugs
* Patients, who the dietician accesses are familiar with low FODMAP diet and therefore is able to identify the placebo diet
* Patients with complicated dietary needs, e.g. severe allergies or intolerances (including lactose and fructose intolerance), athletes, any type of vegetarianism or metabolic diseases
* Pregnancy or planned pregnancy during the study period

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Compliance to the diet measured by a self-administered questionnaire with a percentage scale for every meal consumed | four weeks
How manageable the participants experience the diet, measured by semi-quantitative questionnaire designed by the study group | four weeks
Identification of intervention group measured by the question: "What group do you think you were assigned to?" | four weeks

SECONDARY OUTCOMES:
Gastrointestinal symptoms measured by the questionnaire: The Gastrointestinal symptom rating scale (GSRS) irritable bowel syndrome (IBS) version | four weeks
IBS related quality of life measured by the questionnaire: Irritable bowel syndrome - Quality of Life | four weeks
Endometriosis related quality of life measured by the questionnaire: The Endometriosis Health Profile (EHP-30) | four weeks
Intake of nutrients calculated in by: The Monash University Comprehensive Food Frequency Questionnaire (CNAQ) based on the participants self-reported 7-days food registration | four weeks
Intermenstrual pain measured by VAS scale | four weeks
Global symptom relief measured by the question: "Did you have sufficient relief in your IBS-symptoms during the last 7 days?" | four weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark